CLINICAL TRIAL: NCT02431416
Title: Effect of a GnRH Injection on Ghrelin Concentrations in Girls With Suspected Precocious Puberty
Brief Title: Effect of a GnRH Injection on Ghrelin Concentrations in Girls With Suspected Premature Puberty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Region Örebro County (Other)
Collaborators: Uppsala-Örebro Regional Research Council (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: OLL-430981
Record Dates: First submitted 2015-04-10; First posted 2015-05-01 (Estimated); Last update posted 2019-04-01 (Actual); Status verified 2019-03

CONDITIONS: Puberty, Precocious
Keywords: females; ghrelin; GnRH; randomized, controlled study; children
MeSH Terms: conditions — Puberty, Precocious | interventions — Gonadotropin-Releasing Hormone; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Gonadotropin releasing hormone (GnRH) (Active Comparator): A single intravenous injection of gonadotropin releasing hormone GnRH (Relefact LHRH 0,1 mg/mL). Dose: 100 micrograms per square meter body surface. Maximal dose: 100 micrograms.
  Interventions: Drug: Gonadotropin releasing hormone (GnRH)
- Sodium chloride (Placebo Comparator): A single intravenous injection of sodium chlorid (9 mg/mL). Dose: the same volume as the volume given/to be given with GnRH, that is maximal dose = 1 mL = 9 mg sodium chlorid.
  Interventions: Drug: Sodium Chloride

INTERVENTIONS:
Drug: Gonadotropin releasing hormone (GnRH) — Gonadotropin releasing hormone GnRH (Relefact LHRH) iv injection, single dose, 100 micrograms/square meter body surface, maximum dose: 100 microgram.
  Other Names: Relefact LHRH
  Arms: Gonadotropin releasing hormone (GnRH)
Drug: Sodium Chloride — Sodium chlorid 9 mg/mL will be given as a single iv injection with the same volume as the volume used for the active substance injection.
  Other Names: Saline; placebo
  Arms: Sodium chloride

SUMMARY:
The purposes of the study is to investigate whether circulating levels of ghrelin decreases after an iv injection of GnRH in girls with suspected central premature puberty and to investigate the effects of different post sampling handling on the preservation of acylated ghrelin.

DETAILED DESCRIPTION:
Patients with clinically suspected central premature puberty undergo a GnRH stimulation test to have an appropriate diagnosis. 20 such girls will be recruited to this study and a modified GnRH stimulation test will be done. The modification includes prolonged blood sampling time (0, 30, 60, 90, 120, and 150 min after the GnRH injection instead of the usual 0, 30, 60, and 90 min). The girls will also be investigated twice. In randomised order they will be given either GnRH or placebo (isotone saline), on different days. One week to one month will separate the different investigation days.

The proteinase inhibitor 4-(2-aminoethyl) benzene-sulfonyl fluoride hydrochlorid (AEBSF) will be added to some of the blood tubes, and hydrochloric acid will be added to some of the plasma. All plasma samples will be frozen and all analyses will be done at the same time. Acylated ghrelin will be analyzed by Millipore's specific ELISA kit and deacylated ghrelin will be analyzed by Cayman's specific ELISA kit.

Anthropometric data as well as pubertal state will be collected. P-glucose, S-insulin, S-follicle stimulating hormone (FSH), S-luteinizing hormone (LH), and S-estradiol will also be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Female gender.
* Clinical suspicion of central precocious puberty.
* A GnRH stimulation test is to be performed to make appropriate diagnosis.

Exclusion Criteria:

* Age < 1 year.
* Weight < 10 kg.
* Untreated hypo- or hyperthyroidism.
* Diabetes of any kind.
* BMI > 3 z-score.
* Growth hormone treatment.
* Syndrome or suspected syndrome.
* Tumour or congenital malformation of the hypothalamus or the pituitary gland. (Neuroradiology does not have to be performed only because of the study.)
* On going ulcus ventriculi or the patient has gone through surgery that removed part of the ventricle or changed it markedly in any other way.

Min Age: 1 Year | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
Ghrelin concentration after GnRH injection and after saline injection | 30-150 min after iv injections
  Paired comparison will be done between the acylated ghrelin concentration after GnRH injection and the acylated ghrelin concentration after saline injection.
  Paired comparison will also be done between deacylated ghrelin concentration after GnRH injection and deacylated ghrelin concentration after saline injection.

SECONDARY OUTCOMES:
Deacylated ghrelin concentrations in samples treated with the inhibitor AEBSF, in samples treated with both AEBSF and hydrochloric acid, and in samples not treated with either AEBSF or hydrochloric acid | At baseline
  Concentrations of deacylated ghrelin will be compared between different handling procedures.
Deacylated ghrelin concentrations in samples treated with the inhibitor AEBSF, in samples treated with both AEBSF and hydrochloric acid, and in samples not treated with either AEBSF or hydrochloric acid | 150 min after iv injections
  Deacylated ghrelin concentrations will be compared at 150 min after iv injections between different handling procedures.
Acylated ghrelin concentrations in samples treated with and without hydrochloric acid | 0-150 min after iv injections
  Acylated ghrelin concentrations will be compared between different handling procedures.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Lodefalk, MD, PhD, Principal Investigator — Department of Paediatrics, Faculty of Medicine and Health, Örebro University
Locations (1):
- Department of Paediatrics, Örebro University Hospital, Örebro, Sweden

IPD SHARING:
Plan to Share IPD: No